CLINICAL TRIAL: NCT06330714
Title: Remote Monitoring of Chronic Illness Patients (REMOTE-HUB-1) Study - to Assess Utility of a Mobile Device for Improved Management of At-risk Patients
Brief Title: Remote Monitoring of Chronic Illness Patients With a IHAP Home Wireless Hub and Vitals Measurements
Acronym: REMOTE-HUB-1
Status: Completed | Type: Observational
Sponsor: Aventyn, Inc. (Industry)
Collaborators: Intel Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: AV.RMH.v01-01
Record Dates: First submitted 2018-08-28; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Chronic Disease of Cardiovascular System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Symptoms of chronic illness. — The patient is advised to monitor BP and body weight daily in a standardized fashion as described below:
  * Body weight should be measured in the morning without clothes or shoes after emptying the urinary bladder but before breakfast.
  * BP should be measured in the morning preferably using the right arm, sitting comfortably in a chair after 5 minutes of rest in the seated position.

SUMMARY:
This is planned as a feasibility study.

The primary objective is to evaluate a specially designed patient monitoring software Vitalbeat and standard mobile device hub termed Intel Health Application Platform (IHAP) in terms of its reliability, seamless data transmission and early data availability to the physician to improve patient physician interaction.

The second objective is assessing patient response to use of mobile device monitoring and patient self-monitoring skills to transmit vital signs data using the IHAP wireless home hub device

DETAILED DESCRIPTION:
The proposed study is a prospective single-center clinical feasibility study. All patients shall be monitored for a total period of 30 days from their date of recruitment. A total of 10 patients will be recruited from one center. The center will be provided with mobile devices which would be activated by a local mobile service provider. Additionally a tablet computer will be provided to the local investigator for monitoring patient's data, providing portability and immediate access of information. An automated blood pressure (BP) monitoring apparatus and a weighing scale will be provided to the patient.

Vitalbeat software, with a mobile device home hub having a specially designed patient personalized software application ("Vitalbeat" from Aventyn, USA) for remote monitoring and a clinician monitoring software will be tested in the proposed study. The software has been developed in a manner which provides easy navigation and use, with provision of regular data entry of basic parameters used in chronic illness monitoring. The entered data is instantaneously available on the software monitored at the physician's end.

This study is targeted towards chronic patients. A "chronic" patient is defined as a patient who has had within the last six months symptoms of chronic illness before enrollment.

All patients above 18 years hospitalized and discharged alive with a primary diagnosis of a chronic illness shall be considered for recruitment. Upon enrollment into the study, patients will have mobile device monitoring along with existing standard care monitoring available at the local center.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either gender and 18 years or older
* The subject is able and willing to provide written informed consent prior to enrollment in the study
* Symptoms of chronic illness.

Exclusion Criteria:

* Disability of fingers or upper limbs (unable to use devices)
* Visually impaired
* Those unable to read and write
* Hearing dysfunction
* Significant cognitive disabilities / mental illness
* Those who are unable to handle electronic devices
* Those residing in places outside mobile phone coverage
* Patients who may not come for follow up or likely to drop out of the study
* Any illness which may preclude regular follow up

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study is targeted towards chronic patients. A "chronic" patient is defined as a patient who has had within the last six months symptoms of chronic illness before enrollment.
  All patients above 18 years hospitalized and discharged alive with a primary diagnosis of a chronic illness shall be considered for recruitment. Upon enrollment into the study, patients will have mobile device monitoring along with existing standard care monitoring available at the local center.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Mobile Home Device Hub Data Resiliency | 30 Days
  he primary objective is to evaluate a specially designed patient monitoring software and standard mobile device hub in terms of its reliability, seamless data transmission and early data availability to the physician to improve patient physician interaction once per day for 30 days.

SECONDARY OUTCOMES:
Patient Self Monitoring | 30 Days
  The second objective is assessing patient response to use of mobile device monitoring and patient self-monitoring skills to transmit vital signs data using a home hub device once per day for 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Liver Health, Chandler, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Thorvaldsen T, Benson L, Stahlberg M, Dahlstrom U, Edner M, Lund LH. Triage of patients with moderate to severe heart failure: who should be referred to a heart failure center? J Am Coll Cardiol. 2014 Feb 25;63(7):661-671. doi: 10.1016/j.jacc.2013.10.017. Epub 2013 Oct 30. PMID 24161453
- See also: Assess Measurements of Wireless Cardiac Output Device (Remote-CO-1) — https://clinicaltrials.gov/ct2/show/NCT02252757?term=aventyn&rank=1